CLINICAL TRIAL: NCT04663711
Title: The Degree of Adherence of Pre-anesthetic Tests at Kasr Alaini Hospital to the NICE-Uk Guidelines, and Its Effect on Decision Making & Patient Outcome. Prospective Observational Study
Brief Title: The Degree of Adherence of Pre-anesthetic Tests at Kasr Alaini Hospital to the NICE-Uk Guidelines
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed abdel ghany ali, lecturer of anesthesia, faculty of medicine,Cairo unversity, Cairo University
Other Study IDs: MS-163-2020
Record Dates: First submitted 2020-08-25; First posted 2020-12-11 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Anesthesia
Keywords: preoperative; Investigation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: degree of adherence of pre-anesthetic tests at kasr Alaini hospital to the NICE-Uk guidelines — The anesthesiologist, whom is in charge of preoperative assessment at each unit, will assess patients who are scheduled for elective surgery, and will inform senior anesthesiologists with a minimum 3 years of experience.
  preoperative investigations will be divided into: First part will be on patient's gender, ASA classification, medical history and examination.
  Second part will be on Grade of surgery - Minor/ Intermediate/ Major or complex.
  Third part is requested investigation(s), its rationale, the hierarchy of anesthesiologist requested, and the planned date for surgery.
  Fourth part is about whether that investigation(s) is adherent with NICE-UK guidelines or not.

SUMMARY:
The aim of this study is to assess the effectiveness and usefulness of the current practice of various examinations ordered by anesthesiologists during the pre-anesthetic evaluation in patients who are intended for elective surgery in our hospital. We will also evaluate the effect of delay & its value to predict postoperative complications.

DETAILED DESCRIPTION:
For each preoperative requested test, we will determine whether the test is indicated based on the National Institute for Health and Clinical Excellence (NICE) guidelines and whether it was effective for adverse effects management or unnecessarily requested.

An adherent test was defined as a test that followed NICE, while a non-adherent test was defined as a test that included an over or under test. Normal test results are based on the laboratory reference range of normal values.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients that will be scheduled for an elective general surgical operation during our study time frame.

Exclusion Criteria:

* Patients that are operated on an emergency basis.
* Pregnant females.
* patients scheduled for cardiothoracic and neurosurgical procedures.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients that will be scheduled for an elective general surgical operation during our study time frame
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Percentage of adherence test to NiCE-UK guidelines | 24 hours
  The degree of adherence of the current practices of our institute preoperative testing to the NICE-UK guidelines determined as a percentage

SECONDARY OUTCOMES:
Percentage of overdone investigations | 24 hours
  •The percentage of "overdone" (unnecessary) investigations not recommended by the NICE guidelines which resulted in operative delay & prolonged hospital stay
Estimated cost of overdone investigations | 1 month
  • To assess the impact of requested non recommended investigations by NICE guidelines for preoperative testing on hospital resources (Ordering further investigation - Ordering elective ICU - Increasing hospital stay days)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided